CLINICAL TRIAL: NCT00032383
Title: Complementary/Alternative Medicine for Vestibulopathy
Brief Title: Complementary/Alternative Medicine for Abnormality in the Vestibular (Balance) System
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21AT000553-01 (NIH)
Record Dates: First submitted 2002-03-20; First posted 2002-03-22 (Estimated); Last update posted 2007-01-22 (Estimated); Status verified 2006-07

CONDITIONS: Vestibular Neuronitis; Vestibulopathy
Keywords: Rehabilitation; Tai Chi
MeSH Terms: conditions — Vestibular Neuronitis | interventions — Tai Ji

INTERVENTIONS:
Behavioral: Tai Chi

SUMMARY:
The purpose of this study is to determine the relative merits of vestibular rehabilitation and Tai Chi for patients with inner ear (vestibular) disorders.

DETAILED DESCRIPTION:
It is proposed a randomized, blinded, controlled trial comparing vestibular rehabilitation (VR) to Tai Chi (TC). Our overall goal is to explore whether, and if so, how TC can improve functional, dynamic stability in persons with vestibulopathy (VSP). It is hypothesized that the TC group will demonstrate significantly greater improvement in performing functional activities than the VR group.

Sixty subjects will be randomly assigned into either TC instruction or VR. Both treatment groups will receive identical duration treatment once a week for 10 weeks, with supplemental home exercises. It is hypothesized that 1) TC improves whole-body dynamic locomotor stability more than does VR; 2) TC improves gait coordination during planned and unplanned obstacle encounters more than does VR; 3) TC improves whole-body speed related movement control more than does VR.

ELIGIBILITY:
Main inclusion criteria:

* vestibulopathy and locomotor unsteadiness

Main exclusion criteria:

* diseases/impairments that prevent rehab participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2001-04; Study Completion 2003-04

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital Biomotion Laboratory, Boston, Massachusetts, United States

REFERENCES:
- See also: Click here to visit the Massachusetts General Hospital. — http://www.massgeneral.org/departments.html